CLINICAL TRIAL: NCT05009355
Title: The Effect of Vitamin C Supplementation on GCF Total Oxidant Capacity in Smoker Patients With Periodontitis Following Non-surgical Periodontal Therapy. A Randomized Controlled Clinical Trial
Brief Title: The Effect of Vitamin C on GCF Total Oxidant Capacity in Smoker Patients With Periodontitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer hassan sharafuddin, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100200
Record Dates: First submitted 2021-08-02; First posted 2021-08-17 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Vitamin C Deficiency
MeSH Terms: conditions — Ascorbic Acid Deficiency | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): A Group: Consisted of 20 patients who were treated with scaling and root planing in conjunction with 2g antioxidant Vit (C)
  Interventions: Drug: Vitamin C
- Control (No Intervention): A Group: consisted of 20 patients who were treated with scaling and root planing.

INTERVENTIONS:
Drug: Vitamin C — antioxidant
  Other Names: c retard
  Arms: experimental

SUMMARY:
The effect of vitamin C supplementation on GCF total oxidant capacity in smoker patients with periodontitis following non-surgical periodontal therapy.

DETAILED DESCRIPTION:
All subjects were screened by comprehensive periodontal examination and full periodontal charts were obtained and full-mouth periapical radiographs were taken using the long cone parallel technique at the time of the initial examination to confirm the diagnosis.

Both groups (smokers with stage III-IV grade B periodontitis) received full mouth scaling and root planing using ultrasonic scaler and hand instruments under local anesthesia, completed over 2 visits. Patients were given careful instruction in self performed plaque control measures: twice daily tooth brushing with a brush and tooth paste and once daily interdental cleaning using triangular wooden tooth picks and/or interdental brushes rinsing with 0.125% Chlorhexidine HCL mouthwash (Hexitol® ) to be used twice daily for 2 weeks. Group II received antioxidant vit C 2 grams / day for four weeks.

Collection of gingival crevicular fluid (GCF) sample:

In both groups, GCF samples were collected at the initial visit and collected again 3 months after non-surgical treatment as follows : at the selected area (the most periodontally affected site), all clinically detected supragingival plaque were removed carefully to minimize contamination of the paper strips by the plaque . The teeth selected were then gently washed with water, and the sites under study were isolated with cotton rolls to prevent contamination with saliva and gently dried with an air syringe . Filter paper strips were placed at the entrance of the crevice and were left in place for 30 secs ) and then placed in plastic eppendorf. Strips with any plaque, saliva, or blood contamination were discarded .The sample from the individual site was stored at -80°C for later processing . GCF was then extracted and assayed for the content of total oxidant capacity.

Quantitation of TOC in GCF:

GCF samples of both groups were assayed using ELISA technique for estimation of the level of total oxidant capacity (TOC) in GCF as follows:

The TOC was extracted from the paper strip by adding 100 μl of phosphate buffer saline to the eppendorf tube then mixed by vortex followed by centrifugation for 10 min at 3000Xg. The supernatant was used for estimation of TOC. For the quantitative determination of human TOC concentrations in GCF, PerOx (TOS/TOC) Immun-diagnostik Assay (ELISA) Kit was used. ELISA is intended for the quantitative determination of the total oxidative status/capacity (TOS/TOC) in Ethylene-diaminetetraacetic acid (EDTA)-plasma, serum and cell culture supernatants.

The determination of the peroxides is performed by the reaction of a peroxidase with peroxides in the sample followed by the conversion of TMB (Tetra-methylbenzidine) to a colored product. After addition of a stop solution the samples were measured at 450 nm in a microtiter plate reader. The quantification is performed by the delivered calibrator

ELIGIBILITY:
Inclusion Criteria:

* all patients were systemically healthy
* stage III-IV grade B periodontitis
* A minimum of two non-adjacent teeth having sites with ≥ 5 mm interdental clinical attachment loss .
* Radiographic bone loss extending to middle third of root and beyond .
* All patients were heavy smokers i.e ≥ 20 cigarettes / day .

Exclusion Criteria:

* patients who had received any periodontal or antibiotic treatment or vitamins supplementation during the last six months.
* pregnant or lactating women
* patients who refused to provide written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-12-21 (Estimated)

PRIMARY OUTCOMES:
Total Oxidant Capacity | one month
  unit

SECONDARY OUTCOMES:
Gingival index | one month
  score (0 is good no bleeding 3 is worst spontaneous bleeding )
plaque index | one month
  score (0 is good no plaque 3 is the worst )
probing depth | one month
  mm

CONTACTS AND LOCATIONS:
Overall Officials: abeer H Sharafuddin, PhD, Principal Investigator — Cairo University
Locations (1):
- Abeer Hassan Sharafuddin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No